CLINICAL TRIAL: NCT03902535
Title: Geriatric Assessment and Quality of Life in Older Adults Undergoing Definitive Treatment for Head and Neck or Lung Cancer and Their Informal Caregivers
Brief Title: Geriatric and Quality of Life Assessments in Older Patients With Non-metastatic or Metastatic Head and Neck or Lung Cancer Undergoing Surgery or Chemoradiation and Their Caregivers
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18294; NCI-2018-02024 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18294 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Caregiver; Head and Neck Carcinoma; Lung Carcinoma; Metastatic Head and Neck Carcinoma; Metastatic Lung Carcinoma; Stage 0 Lung Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (geriatric and quality of life assessments): Patients complete comprehensive geriatric and quality of life assessments within 1-4 weeks of treatment (either upfront surgery which may be followed by radiation with or without chemotherapy or upfront radiation which may include CRT) initiation (baseline), and at 1, 3, and 6 months following CRT completion.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (quality of life assessment): Family caregivers complete quality of life assessment at baseline, and at 1, 3, and 6 months following patient radiation or CRT completion.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Complete comprehensive geriatric assessment
  Groups: Group I (geriatric and quality of life assessments)
Other: Quality-of-Life Assessment — Complete quality of life assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies comprehensive geriatric and quality of life assessments in older patients with head and neck or lung cancer that has or has not spread to other parts of the body who are undergoing standard surgery or chemoradiation, and their caregivers. Comprehensive geriatric assessment may improve the quality of life of patients with head and neck or lung cancer and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the patterns and distribution of comprehensive geriatric assessment (CGA) scores and physical activity levels and quality of life measures in older (>= 65) patients with non-metastatic or metastatic head and neck or lung cancer undergoing upfront surgery followed (may be followed by adjuvant therapy) or upfront definitive radiation (with or without chemotherapy at the same time) to cure the disease.

II. To describe the incidence and type of grade 2-5 toxicities in this patient population.

III. To describe the family caregiver (FCG)-reported caregiving burden level and quality of life (QOL) scores.

SECONDARY OBJECTIVES:

I. To identify areas of vulnerability in this patient population using the geriatric assessment.

II. To identify potential referrals based on geriatric assessment results. III. To describe other healthcare resource use and potential treatment modifications (unplanned hospitalization, emergency room (ER) visits, readmission rates, breaks in radiation and/or chemoradiation (CRT), dose modifications).

IV. To explore changes in geriatric assessment and patient-reported symptoms, QOL, weight, and functional status from pre-treatment to 3-months, 6 months post-treatment.

V. To explore changes in family caregiver (FCG)-reported caregiving burden and QOL from pre-treatment to 3-months, 6 months post-treatment.

VI. To explore the relationship between geriatric assessment results and patient-reported symptoms and QOL.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Patients complete comprehensive geriatric and quality of life assessments within 1-4 weeks of treatment (either upfront surgery which may be followed by radiation with or without chemotherapy or upfront radiation which may include CRT) initiation (baseline), and at 1, 3, and 6 months following CRT completion.

GROUP II: Family caregivers complete quality of life assessment at baseline, and at 1, 3, and 6 months following patient radiation or CRT completion.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Diagnosed with non-metastatic or metastatic head and neck cancer or lung cancer
* PATIENT: Scheduled to undergo either upfront surgery or definitive radiation treatment (including CRT)
* PATIENT: Age >= 65 years
* PATIENT: Able to read and understand English
* FAMILY CAREGIVER: Family member/friend identified by the patient as the primary caregiver before and after surgery and/or radiation (including CRT)
* FAMILY CAREGIVER: Age >= 21 years
* FAMILY CAREGIVER: Able to read and understand English
* ALL SUBJECTS: Must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo upfront surgery or concurrent CRT for non-metastatic head and neck cancer and family caregivers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Comprehensive geriatric assessment (CGA) scores and domains | Up to 6 months post therapy
  Descriptive statistics will be used to summarize all CGA measure scores/domains.
Physical activity levels | Up to 6 months post therapy
  Descriptive statistics will be used to summarize all physical activity levels.
Quality of life (QOL) measures | Up to 6 months post therapy
  Descriptive statistics will be used to summarize all QOL measures.
Incidence and type of grade 2-5 toxicities | Up to week 4
  Types of grade 2-5 toxicities will be summarized and proportions of patients with grade 2-5 toxicities will be tabulated and reported according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Family caregiver (FCG)-reported caregiving burden level and QOL scores | Up to 6 months post therapy
  Descriptive statistics will be used to summarize all FCG-reported measure scores/domains.

SECONDARY OUTCOMES:
Percentage of patients with vulnerability using the geriatric assessment | Up to 6 months post therapy
  Percentage of patients with vulnerability will be calculated as the number of patients with vulnerability divided by 30 (target sample).
Percentage of patients who receive and accept referrals | Up to 6 months post therapy
  The percentage of patients who receive and accept referrals will be calculated as the number of patients with referral divided by the number of patients with vulnerability.
Treatment modification and healthcare utilization in patients | Up to week 12
  Frequency and reasons for healthcare resource use and treatment modifications will be tabulated.
Change in CGA scores and domains | Baseline up to 6 months post therapy
  Changes will be calculated as post-treatment scores minus pre-treatment scores. The pattern of changes in CGA assessment will be summarized.
Change in physical activity levels | Baseline up to 6 months post therapy
  Will utilize the pedometer to assess physical activity level during and after treatment and record changes. The pattern of changes in physical activity levels will be summarized.
Change in QOL measures | Baseline up to 6 months post therapy
  Changes will be calculated as post-treatment scores minus pre-treatment scores. The pattern of changes in QOL measures will be summarized.
Change in FCG-reported caregiving burden level and QOL scores | Baseline up to 6 months post therapy
  Changes will be calculated as post-treatment scores minus pre-treatment scores.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States